CLINICAL TRIAL: NCT00712868
Title: Safety Dermatological Evaluation: Acceptability With Gynaecological Follow up Lactacyd Femina
Brief Title: Acceptability of Lactacyd Femina
Acronym: LACTAFEM
Status: Completed | Phase: Phase 4 | Type: Interventional
Sponsor: Sanofi (Industry)
Responsible Party: Medical Affairs Study Director, sanofi-aventis
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: LACAC_L_03447
Record Dates: First submitted 2008-07-07; First posted 2008-07-10 (Estimated); Last update posted 2009-07-20 (Estimated); Status verified 2009-07

CONDITIONS: Hygiene
MeSH Terms: interventions — Lactic Acid

ARMS (1):
- 1 (Experimental): Lactic Acid once a day during 21 days
  Interventions: Drug: Lactic acid

INTERVENTIONS:
Drug: Lactic acid — Once a day

SUMMARY:
To demonstrate the safety and acceptability of the gynaecological formulation.

ELIGIBILITY:
Inclusion Criteria:

* Integral skin in the tested region

Exclusion Criteria:

* Pregnancy or breastfeeding women
* Use of anti-inflammatory or immune-suppression drugs
* Topical medication use at the tested region
* Active cutaneous gynaecological disease which may interfere in study results
* Personal history of allergic disease at the area to be treated
* Allergic or atopic history

The above information is not intended to contain all considerations relevant to a patient's potential participation in a clinical trial.

Ages: 18 Years to 60 Years | Sex: Female | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 559 (Actual)
Dates: Start 2008-06; Primary Completion 2008-08 (Actual); Study Completion 2008-08 (Actual)

PRIMARY OUTCOMES:
Clinical and local tolerability | After 21 days

CONTACTS AND LOCATIONS:
Overall Officials: Judith Diaz, Md, Study Director — Sanofi
Locations (1):
- Sanofi-Aventis Administrative Office, Col. Coyoacan, Mexico